CLINICAL TRIAL: NCT04145037
Title: The Guard1 Trial, an Open-Label, Multinational Phase 1/2 Study of the Safety and Efficacy of Ex Vivo, Lentiviral Vector-Mediated Gene Therapy AVR-RD-02 for Subjects With Type 1 Gaucher Disease
Brief Title: Lentiviral Vector Gene Therapy - The Guard1 Trial of AVR-RD-02 for Subjects With Type 1 Gaucher Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This study was voluntarily terminated by the sponsor to halt development and was not based on any safety or medical reasons.
Sponsor: AVROBIO (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVRO-RD-02-201
Record Dates: First submitted 2019-08-27; First posted 2019-10-30 (Actual); Results first posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-10

CONDITIONS: Gaucher Disease
Keywords: Type 1 Gaucher; Guard1
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Switch Stable (Experimental): Switch-stable arm: Subjects who had undergone ERT ≥15 U/kg and ≤60 U/kg every other week (or equivalent; i.e., any combination of infusions resulting in a total monthly ERT dose of >30 U/kg and <120 U/kg) for ≥24 consecutive months for Type 1 Gaucher disease at the time of Screening. Switch-stable subjects must have discontinued ERT at least 2 weeks before the scheduled AVR-RD-02 infusion. Switch-stable subjects who had been and substrate reduction therapy (SRT) must not have received SRT within 12 months of Screening.
  Interventions: Drug: AVR-RD-02
- Treatment-naïve (Experimental): Treatment-naïve arm: Subjects with Type 1 Gaucher disease who had never received either ERT or SRT for Gaucher disease or had not received either ERT or SRT for Gaucher disease within 12 months of Screening (i.e., treatment-naïve subjects). Enrollment followed a similar scheme as for the switch-stable subjects.
  Note: No subjects enrolled in this arm.
  Interventions: Drug: AVR-RD-02

INTERVENTIONS:
Drug: AVR-RD-02 — AVR-RD-02 Drug product: active substance is autologous CD34+ enriched hematopoietic stem cells (HSCs) that have been genetically modified ex vivo with a lentiviral vector (LV) to contain a ribonucleic acid (RNA) transcript that, after reverse transcription, results in codon-optimized, complementary deoxyribonucleic acid (cDNA) that, upon its integration into human genome, encodes for functional human glucocerebrosidase (GCase).

SUMMARY:
This was a multinational, open-label study to assess the safety and efficacy of AVR-RD-02 in approximately 8 to 16 subjects (male or female) who are ≥18 and ≤50 years of age and post pubertal at Screening with a confirmed diagnosis of Type 1 Gaucher disease (based on clinical phenotype, genotyping, and deficient GCase enzyme activity in whole blood).

DETAILED DESCRIPTION:
Five study periods (Screening, Baseline, Pre-gene Therapy Infusion, Gene Therapy Infusion, and Post-gene Therapy Infusion Follow-up) comprised the study. During the Screening Period (approximately 60 days), written informed consent was obtained and the subject completed other Screening procedures to confirm study eligibility. Once study eligibility was confirmed, subjects entered the Baseline Period (up to 7 days) during which time assessments were performed to establish Pre-gene Therapy Infusion baseline. Once baseline assessments were completed, the subject entered the Pre-gene Therapy Infusion Period (approximately 8 to 10 weeks) during which time mobilization, apheresis, AVR-RD-02 investigational product preparation and testing for release, busulfan conditioning regimen administration took place. Enzyme replacement therapy was discontinued at least 2 weeks before the scheduled Gene Therapy Infusion Day. Following completion of the Pre-gene Therapy Infusion Period, the subject entered the Gene Therapy Infusion Period (1 day) during which AVR-RD-02 infusion took place. After AVR-RD-02 Gene Therapy Infusion, the subject entered the Post-gene Therapy Infusion Follow-up Period (approximately 52 weeks) during which time periodic safety and efficacy assessments were performed to assess measures of safety, engraftment, and clinical response following AV-RD-02 infusion.

In August 2023, the study was terminated early by the Sponsor, which was not based on any safety or medical reasons and therefore, one subject did not complete the study (i.e., Week 52). Subsequently, in August 2023, the sponsor's long-term follow-up study (AVRO-RD-02-LTF01), was also terminated early for the same reason as the AVRO-RD-02-201 study, and therefore, no subjects completed the 15-year long-term follow-up study.

ELIGIBILITY:
INCLUSION CRITERIA for all Enrolled (Switch-stable and Treatment-naïve) Subjects:

Note: No treatment-naïve subjects enrolled in this study.

1. Subject was ≥18 and ≤50 years old and post pubertal
2. Subject had a confirmed diagnosis of Type 1 Gaucher disease based on deficient GCase enzyme at Screening.

   a. For switch-stable subjects, documentation of GCase enzyme activity prior to having been started on ERT or if GCase levels prior to ERT were not available, deficient trough GCase enzyme activity in peripheral blood at Screening.
3. Female subjects of reproductive potential were counseled regarding the risks, benefits, limitations, and alternatives associated with female fertility preservation. Oocyte harvesting and cryopreservation were offered
4. Male subjects were willing to refrain from donating sperm at any time after receiving conditioning therapy. For subjects planning on (or for whom there is a possibility of) fathering children in the future, sperm cryopreservation before administration of the conditioning regimen was recommended.
5. All subjects who had not undergone successful surgical sterilization (ie, vasectomy, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) agreed to remain sexually abstinent or use two effective methods of contraception while sexually active from the day of conditioning administration until 52 weeks post-gene therapy infusion. Two methods of contraception were required even with documented medical assessment of surgical success of sterilization.

   1. For male subjects and for male spouses/partners of female subjects, condoms were an acceptable method of barrier contraception
   2. For female subjects and for female spouses/partners of male subjects, acceptable methods of barrier contraception included diaphragm, cervical cap, or contraceptive sponge.
6. Male and female subjects agreed to refrain from donating sperm and eggs, respectively, after undergoing conditioning.
7. Subject was willing to refrain from donating blood, organs, tissues, or cells for gene therapy infusion any time after AVR-RD-02 treatment.
8. Subject was willing and able to provide written informed consent for the study in accordance with applicable regulations and guidelines and to comply with all study visits and procedures, including the use of any data collection device(s) that may be used to directly record subject data.
9. Subject was willing to receive blood or blood products transfusion to manage adverse events (AEs).

   Additional Inclusion Criteria for Switch-stable Subjects (in addition to criteria 1-9 above):
10. Subject had undergone a stable dose (within 75% to125% of the prescribed dose) of ERT ≥ 15 U/kg and ≤ 60 U/kg every other week (or equivalent) for ≥ 24 consecutive months with no significant interruptions, in dosing over the last 6 months, in the opinion of the Investigator, prior to Screening
11. Subject had normal or near-normal hematologic values at Screening defined as one or more of the following:

    1. Hemoglobin concentration ≥10 g/dL
    2. Platelet count ≥80 x 10^9/L
12. Subject had stable Gaucher disease during the 6 months immediately preceding Screening defined by:

    1. Stable hemoglobin concentration (i.e., within a range of ±2 g/dL of the Screening value) based on documented historical clinical laboratory results and
    2. Stable platelet count (within ±20% of the Screening value) based on documented historical clinical laboratory results
13. Subject had not received SRT for Gaucher disease within 12 months of Screening

    Additional Inclusion Criteria for Treatment-naïve Subjects (in addition to inclusion criteria 1 through 9, above, treatment-naïve subjects must meet the following inclusion criteria for participation in this study):
14. Subject had neither received ERT nor SRT for Gaucher disease nor has received neither ERT nor SRT for Gaucher disease within 12 months of Screening.
15. Subject had a hemoglobin level ≤2 g/dL below the lower limit of normal (LLN) for age and sex at Screening and at least one of the following at Screening:

    1. Platelet count <120 x 10^9/L
    2. Enlarged liver by palpation, confirmed on abdominal MRI
    3. Moderate splenomegaly by palpation, confirmed on abdominal MRI
16. For any subject who was treatment-naïve, ERT peri-procedurally (from the Screening Period throughout 2 weeks prior to Gene Therapy Infusion) was considered in consultation with the PI and Sponsor Medical Monitor.

EXCLUSION CRITERIA:

1. Subject had Type 2 or 3 Gaucher disease, had severe neurological signs and symptoms, defined as complete ocular paralysis, overt myoclonus or history of seizures, characteristic of neuronopathic Gaucher disease, or had a tremor, peripheral neuropathy or symptoms of Parkinson's disease.

Subject had any one of the following:

1. Hemoglobin value <9.0 g/dL, or
2. Platelet count <70 x 10˄9/L, or
3. Spleen volume >10 x normal, or
4. Pulmonary hypertension 3. Subject had experienced a prior anaphylactic or anaphylactoid reaction (of any severity) to ERT.

   4. Treatment-naïve subject had history of clinically significant (CS) anti-GCase antibodies.

   5. Subject had a contraindication to ERT, in the opinion of the Investigator. 6. Subject had a contraindication to HSC transplantation (HSCT), in the opinion of the Investigator.

   7. Subject presented with iron, folic acid, and/or vitamin B12 deficiency sustained anemia during Screening.

   8. Subject had idiopathic thrombocytopenic purpura (ITP), thrombotic thrombocytopenic purpura (TTP), thrombocytopenia, anemia, hepatomegaly, splenomegaly, and/or osteoporosis, unrelated to Gaucher disease, in the opinion of the Investigator.

   9. Subject had a clinical co-morbidity such as neurologic, cardiovascular, pulmonary, hepatic, gastrointestinal, renal, hematologic, endocrine, metabolic, genetic, immunologic, neoplastic, or psychiatric disease, other medical condition(s), or intercurrent illnesses that may have confounded the study results or, in the opinion of the Investigator, may have precluded participation in the study.

   10. Subject was a pregnant and/or lactating female. 11. Subject was unable to understand the nature, scope, and possible consequences of the study.

   12. Subject had diabetes mellitus (Type 1 or Type 2). 13. Subject had active, progressive bone necrosis. 14. Subject had an active chronic infection during the Screening, Baseline, or Pre-gene Therapy Infusion Period of the study.

   15. Subject had an active uncontrolled acute bacterial, viral, fungal, parasitic, or prion-associated infection during the Screening, Baseline, or Pre-gene Therapy Infusion Period of the study.

   16. Subject had a history of (or current) tuberculosis. 17. Subject tested positive for hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV, Type 1 or 2), human T-cell lymphotropic virus (HTLV)-1, HTLV-2, and/or syphilis on Venereal Disease Research Laboratory (VDRL) test, chemiluminescent microplate immunoassay (CMIA), or enzyme immunosorbent assay (EIA) at Screening.

   18. Subject had a prior history of (or current) cancer or precancerous lesion or has a known genetic predisposition to cancer. The one exception was a prior history of resected squamous cell carcinoma.

   19. Subject had any other medical condition that predisposes him/her to (or conveys increased risk of) malignancy, in the opinion of the Investigator - including history of (or current) monoclonal gammopathy of undetermined significance (MGUS).

   20. Subject had a history of alcohol or illicit drug abuse, according to the Investigator's judgment.

   21. Subject had undergone, or was scheduled to undergo, bone marrow transplant, HSC transplant, and/or solid organ transplant. NOTE: Subjects who were otherwise eligible for the study but were scheduled for bone marrow or HSC transplant to treat Type 1 Gaucher disease may have been enrolled in the study (instead of receiving an allogeneic transplant) and undergo gene therapy infusion with AVR-RD-02.

   22. Subject had white blood cell count (WBC) < 3.0 x 10˄9/L and/or uncorrected bleeding disorder from enrollment (i.e., signing of informed consent at Screening) through the Gene Therapy Infusion Period of the study (i.e., the day of AVR-RD-02 gene therapy infusion).

   23. Subject had clinically significant immunosuppressive disease or condition, in the opinion of the Investigator, at Screening.

   24. Subject was on (or requires treatment with) cytotoxic or immunosuppressive agents from 60 days prior to signing informed consent at Screening (i.e., study enrollment) through the Week 52 study visit; the one exception was treatment with cytotoxic or immunosuppressive agents required per protocol for stem cell transplant.

   25. Subject was on (or requires treatment with) red blood cell (RBC) growth factor (e.g., erythropoietin) from 6 months prior to enrollment (i.e., signing of informed consent at Screening) through the Week 52 study visit.

   26. Subject had any condition that made it impossible to perform MRI studies. 27. Subject had medical condition(s) and/or was receiving medication(s) that would contraindicate ability to undergo mobilization (including contraindication to granulocyte colony-stimulating factor (G-CSF) and/or plerixafor), apheresis, or conditioning.

   28. Busulfan was contraindicated for the subject. 29. Subject had previously received treatment with AVR-RD-02 or any other gene therapy.

   30. Subject was participating in (or plans to participate in) any other investigational drug trial or plans to be exposed to any other investigational agent, device and/or procedure, from 30 days prior to enrollment (i.e., signing of informed consent at Screening) through study completion.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milena Veselinovic, MD, Study Director — AVROBIO
Locations (5):
- United States (4):
  - University of California San Diego, San Diego, California
  - University of Iowa, Iowa City, Iowa
  - Hackensack University Medical Center, Hackensack, New Jersey
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Switch Stable: Switch-stable arm: Subjects who had undergone ERT ≥15 U/kg and ≤60 U/kg every other week (or equivalent; i.e, any combination of infusions resulting in a total monthly ERT do.se of >30 U/kg and <120 U/kg) for ≥24 consecutive months for Type 1 Gaucher disease at the time of Screening. Switch-stable subjects must have discontinued ERT at least 2 weeks before the scheduled transplant day. Switch-stable subjects who had been on substrate reduction therapy (SRT) must not have received SRT within 12 months of Screening.
  AVR-RD-02: AVR-RD-02 Drug product: active substance is autologous CD34+ enriched hematopoietic stem cells (HSCs) that have been genetically modified ex vivo with a lentiviral vector (LV) to contain a ribonucleic acid (RNA) transcript that, after reverse transcription, results in codon-optimized, complementary deoxyribonucleic acid (cDNA) that, upon its integration into human genome, encodes for functional human glucocerebrosidase (GCase).
- Treatment-naïve: Treatment-naïve arm: Subjects with Type 1 Gaucher disease who had never received either ERT or SRT for Gaucher disease or had not received either ERT or SRT for Gaucher disease within 12 months of Screening (i.e., treatment-naïve subjects). Enrollment followed a similar scheme as for the switch-stable subjects.
  Note : No subjects enrolled in this arm.
  AVR-RD-02: AVR-RD-02 Drug product: active substance is autologous CD34+ enriched hematopoietic stem cells (HSCs) that have been genetically modified ex vivo with a lentiviral vector (LV) to contain a ribonucleic acid (RNA) transcript that, after reverse transcription, results in codon-optimized, complementary deoxyribonucleic acid (cDNA) that, upon its integration into human genome, encodes for functional human glucocerebrosidase (GCase).
Period: Overall Study
Arm/Group | Switch Stable | Treatment-naïve
Started | 8 | 0
Mobilized and Apheresed | 6 | 0
Received AVR-RD-02 | 5 | 0
Completed | 4 | 0
Not Completed | 4 | 0
Not completed — Study terminated | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treatment-naïve arm did not enroll any subjects at the time of study termination.
Groups:
- Switch Stable: Switch-stable arm: Subjects who had undergone ERT ≥15 U/kg and ≤60 U/kg every other week (or equivalent; i.e., any combination of infusions resulting in a total monthly ERT do.se of >30 U/kg and <120 U/kg) for ≥24 consecutive months for Type 1 Gaucher disease at the time of Screening. Switch-stable subjects must have discontinued ERT at least 2 weeks before the scheduled transplant day. Switch-stable subjects who had been on substrate reduction therapy (SRT) must not have received SRT within 12 months of Screening.
  AVR-RD-02: AVR-RD-02 Drug product: active substance is autologous CD34+ enriched hematopoietic stem cells (HSCs) that have been genetically modified ex vivo with a lentiviral vector (LV) to contain a ribonucleic acid (RNA) transcript that, after reverse transcription, results in codon-optimized, complementary deoxyribonucleic acid (cDNA) that, upon its integration into human genome, encodes for functional human glucocerebrosidase (GCase).
- Total: Total of all reporting groups
Arm/Group | Switch Stable | Treatment-naïve | Total
Number analyzed (Participants) | 8 | 0 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 0 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.25 (6.30) |  | 34.25 (6.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 4 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 7 | 0 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 0 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Clinically Significant Adverse Events (AEs) and Serious Adverse Events (SAEs) of AVR-RD-02
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The AE/SAE are also inclusive of any abnormalities in Clinical Laboratory Tests, Vital Signs and in Electrocardiographs (ECGs).
  AE/SAE can either be related to AVR-RD-02 infusion or attributed to the conditioning agent, mobilization agent(s), study procedures, and the underlying disease.
Time Frame: Baseline to 52 weeks post-AVR-RD-02 treatment follow-up
Population: Population consists of switch-stable subjects. Treatment-naïve arm did not enroll any subjects at the time of study termination.
Measure: Number; unit: Number of events
Groups:
- Switch Stable: Switch-stable arm: Subjects who had undergone ERT ≥15 U/kg and ≤60 U/kg every other week (or equivalent; i.e, any combination of infusions resulting in a total monthly ERT dose of >30 U/kg and <120 U/kg) for ≥24 consecutive months for Type 1 Gaucher disease at the time of Screening. Switch-stable subjects must have discontinued ERT at least 2 weeks before the scheduled transplant day. Switch-stable subjects who had been on substrate reduction therapy (SRT) must not have received SRT within 12 months of Screening.
  AVR-RD-02: AVR-RD-02 Drug product: active substance is autologous CD34+ enriched hematopoietic stem cells (HSCs) that have been genetically modified ex vivo with a lentiviral vector (LV) to contain a ribonucleic acid (RNA) transcript that, after reverse transcription, results in codon-optimized, complementary deoxyribonucleic acid (cDNA) that, upon its integration into human genome, encodes for functional human glucocerebrosidase (GCase).
Arm/Group | Switch Stable | Treatment-naïve
Number analyzed (Participants) | 6 | 0
Number of events
  SAEs Related to AVR-RD-02 Infusion | 0 |
  AEs Related to AVR-RD-02 Infusion | 0 |
  SAEs Not Related to AVR-RD-02 Infusion | 2 |
  AEs Not Related to AVR-RD-02 Infusion | 189 |

2. Primary Outcome: Vector Copy Number (VCN) in Peripheral Blood as Assessed by Quantitative Polymerase Chain Reaction (qPCR) and/or Droplet Digital Polymerase Chain Reaction (ddPCR)
Description: VCN, defined as the average number of copies of the therapeutic gene (transgene) in a sample of cells, is conventionally reported as the number of vector copies found in a sample, relative to copies of a reference gene in the human genome. This is an estimate of the number of integration sites per cell (on average). A VCN of 1 would signify that a sample of cells evaluated contains on average at least one [working] copy of the therapeutic transgene per cell. This measurement was for VCN in a sample of progenitor cells obtained from a peripheral blood sample.
Time Frame: Baseline to 52 weeks post-AVR-RD-02 treatment follow-up
Population: as for outcome 1
Measure: Mean (Full Range); unit: number of copies/cell
Arm/Group | Switch Stable | Treatment-naïve
Number analyzed (Participants) | 4 | 0
number of copies/cell | 0.55 [0.17 to 0.86] |

3. Primary Outcome: Vector Copy Number (VCN) in Bone Marrow as Assessed by Quantitative Polymerase Chain Reaction (qPCR) and/or Droplet Digital Polymerase Chain Reaction (ddPCR)
Description: VCN is defined as the average number of copies of the therapeutic gene (transgene) in a sample of cells and is a measurement of the number of copies of the vector found in a sample, relative to copies of a reference gene in the human genome. This is an estimate of the number of integration sites per cell (on average). A VCN of 1 would signify that a sample of cells evaluated contains on average at least one [working] copy of the therapeutic transgene per cell. This measurement was for VCN in a sample of bone marrow progenitor cells obtained from an aspirate.
Time Frame: Baseline to 52 weeks post-AVR-RD-02 treatment follow-up
Population: Population consists of switch-stable subjects. Bone marrow samples were collected and batched for analysis, but due to the early termination of the study, samples were not analyzed and subsequently discarded. Refer to "Limitations and Caveats" section. Treatment-naïve arm did not enroll any subjects at the time of study termination.
Arm/Group | Switch Stable | Treatment-naïve
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Change From Baseline in Spleen Volume Assessed by Abdominal MRI
Description: Percent change in spleen volume = ([spleen volume at Week 52 minus spleen volume at baseline] divided by [spleen volume at baseline]) multiplied by 100. A reduction in the percent change from baseline (%CFB) in spleen volume (mL) is a positive indicator of efficacy.
Time Frame: Baseline to 52 weeks post-AVR-RD-02 treatment follow-up
Population: Population consists of switch-stable subjects. Of the four participants who completed the study, one participant had been splenectomized. Treatment-naïve arm did not enroll any subjects at the time of study termination.
Measure: Mean (Full Range); unit: percentage
Arm/Group | Switch Stable | Treatment-naïve
Number analyzed (Participants) | 3 | 0
percentage | -17.03 [-22.8 to -10.9] |

5. Primary Outcome: Change From Baseline in Liver Volume Assessed by Abdominal MRI
Description: Percent change in liver volume = ([liver volume at Week 52 minus liver volume at baseline] divided by [liver volume at baseline]) multiplied by 100. A reduction in the percent change from baseline (%CFB) in liver volume (mL) is a positive indicator of efficacy.
Time Frame: Baseline to 52 weeks post-AVR-RD-02 treatment follow-up
Population: as for outcome 1
Measure: Mean (Full Range); unit: percentage
Arm/Group | Switch Stable | Treatment-naïve
Number analyzed (Participants) | 4 | 0
percentage | -4.95 [-21.1 to 7.8] |

6. Primary Outcome: Change From Baseline in Hemoglobin Concentration
Description: Ratio to baseline indicates the percent change in hemoglobin concentration. The baseline value is defined as 1 or 100%. A ratio to Baseline <1 indicates a reduction in hemoglobin concentration and a ratio to Baseline >1 indicates an increase in hemoglobin concentration.
Time Frame: Baseline to 52 weeks post-AVR-RD-02 treatment follow-up
Population: as for outcome 1
Measure: Mean (Full Range); unit: ratio
Arm/Group | Switch Stable | Treatment-naïve
Number analyzed (Participants) | 4 | 0
ratio | 1.00 [0.87 to 1.14] |

7. Primary Outcome: Change From Baseline in Platelet Count
Description: Ratio to baseline indicates the percent change in platelet count. The Baseline value is defined as 1 or 100%. A ratio to Baseline <1 indicates a reduction in platelet count and a ratio to Baseline >1 indicates an increase in platelet count.
Time Frame: Baseline to 52 weeks post-AVR-RD-02 treatment follow-up
Population: as for outcome 1
Measure: Mean (Full Range); unit: ratio
Arm/Group | Switch Stable | Treatment-naïve
Number analyzed (Participants) | 4 | 0
ratio | 0.83 [0.64 to 1.08] |

8. Primary Outcome: Change From Baseline in Plasma Lyso-Gb1 Levels by Liquid Chromatography Tandem Mass Spectrometry (LC/MS/MS)
Description: Glucosylsphingosine (lyso-Gb1) is the substrate that accumulates in the lysosomes of patients affected by Gaucher disease as a result of deficiencies in GCase enzyme activity. Treatment with AVR-RD-02 is intended to replace the missing GCase enzymatic activity, which allows degradation of accumulated lyso-Gb1 substrate in the lysosomes. Negative values (decrease from Baseline) are an indicator of efficacy.
Time Frame: Baseline to 52 weeks post-AVR-RD-02 treatment follow-up
Population: as for outcome 1
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Switch Stable | Treatment-naïve
Number analyzed (Participants) | 4 | 0
ng/mL | -12.03 [-29.50 to -0.50] |

9. Secondary Outcome: Change From Baseline in GCase Enzyme Activity Level in Plasma
Description: Treatment-naïve Gaucher patients are deficient in glucosylcerebrosidase (GCase) enzyme activity due to mutations in the GBA gene. AVR-RD-02 is intended to increase the amount of GCase enzyme activity in the lysosomes of treated subjects. A positive value (increase from Baseline in GCase enzyme activity) is a positive indicator of efficacy.
Time Frame: Weeks 13, 26, 39, and 52
Population: as for outcome 1
Measure: Mean (Full Range); unit: μmol/L/h
Arm/Group | Switch Stable | Treatment-naïve
Number analyzed (Participants) | 4 | 0
μmol/L/h
  Week 13 | 7.6 [1.8 to 10.9] |
  Week 26 | 5.0 [4.0 to 5.9] |
  Week 39 | 4.9 [1.7 to 8.4] |
  Week 52 | 1.5 [-1.8 to 3.6] |

10. Secondary Outcome: Change From Baseline in GCase Enzyme Activity Level in Peripheral Blood Leukocytes
Description: as for outcome 9
Time Frame: Weeks 13, 26, 39, and 52
Population: Population consists of switch-stable subjects. Although samples were collected, GCase PBL results were not available at many timepoints due to sample instability, and therefore, only available results are reported in the table below. Refer to "Limitations and Caveats" section. Treatment-naïve arm did not enroll any subjects at the time of study termination
Measure: Mean (Full Range); unit: μmol/g protein/h
Groups:
- Treatment-naïve: Treatment-naïve arm: Subjects with Type 1 Gaucher disease who had never received either ERT or SRT for Gaucher disease or had not received either ERT or SRT for Gaucher disease within 12 months of Screening (i.e., treatment-naïve subjects). Enrollment followed a similar scheme as for the switch-stable subjects.
  Note: No subjects enrolled in this arm.
  AVR-RD-02: AVR-RD-02 Drug product: active substance is autologous CD34+ enriched hematopoietic stem cells (HSCs) that have been genetically modified ex vivo with a lentiviral vector (LV) to contain a ribonucleic acid (RNA) transcript that, after reverse transcription, results in codon-optimized, complementary deoxyribonucleic acid (cDNA) that, upon its integration into human genome, encodes for functional human glucocerebrosidase (GCase).
Arm/Group | Switch Stable | Treatment-naïve
Number analyzed (Participants) | 4 | 0
μmol/g protein/h
  Week 13: number analyzed (Participants) | 2 | 0
  Week 13 | 13.3 [11.0 to 15.6] |
  Week 26: number analyzed (Participants) | 1 | 0
  Week 26 | 19.2 [19.2 to 19.2] |
  Week 39: number analyzed (Participants) | 3 | 0
  Week 39 | 6.0 [0.6 to 13.2] |
  Week 52: number analyzed (Participants) | 3 | 0
  Week 52 | 7.1 [0.2 to 11.5] |

11. Secondary Outcome: Number of Subjects Who Restarted ERT
Description: The absence of the need to re-start ERT post treatment is a positive indicator of efficacy.
Time Frame: Between Week 26 and Week 52 post-AVR-RD-02 treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Switch Stable | Treatment-naïve
Number analyzed (Participants) | 5 | 0
Participants | 0 |

12. Secondary Outcome: Change From Baseline in Presence of Anti-GCase Total Antibodies
Description: Number of subjects with changes in anti-GCase antibodies from Baseline to post infusion timepoints. Unit of measure: Number of subjects negative at baseline but positive at post-treatment timepoints. A negative or zero result (titer lower or unchanged at post-infusion timepoints compared to Baseline) indicates no immune response to the therapeutic protein.
Time Frame: At Weeks 5, 13, 26, 39, and 52
Population: Population consists of switch-stable subjects. One of the five subjects had pre-existing antibodies to GCase due to ERT exposure. This subject had a positive and unchanged low titer at all pre-infusion and post-infusion timepoints. Treatment-naïve arm did not enroll at the time of study termination
Measure: Count of Participants; unit: Participants
Arm/Group | Switch Stable | Treatment-naïve
Number analyzed (Participants) | 5 | 0
Participants
  Week 5 | 0 |
  Week 13 | 0 |
  Week 26 | 0 |
  Week 39 | 0 |
  Week 52 | 0 |

13. Secondary Outcome: Change From Baseline in Bone Mineral Density (BMD) Assessed by Bone Density Scan (DXA)
Description: An increase in BMD is a positive indicator of efficacy. Subjects had T-scores reported for change from baseline in Bone Mineral Density in the Femoral Neck and Lumbar Spine regions assessed by Bone Mineral Density (DXA).
  The T-score on the subject's bone density report shows how many standard deviations the subject's bone mass differs from the bone mass of an average healthy 30-year-old adult. If the bones are more dense than the average 30-year-old adult, the bone mass will be indicated as a positive T-score. Higher positive T-score indicates greater bone density. If the bones are less dense than the average 30-year-old adult, the bone mass will be indicated as a negative T-score. Lower negative T-score indicates lesser bone density.
Time Frame: Baseline to 52 weeks post-AVR-RD-02 treatment follow-up
Population: Population consists of switch-stable subjects. Some subjects had missing baseline and/or Week 52 data, and therefore change from baseline could not be calculated.
  Refer to "Limitations and Caveats" section. Treatment-naïve arm did not enroll any subjects at the time of study termination.
Measure: Mean (Full Range); unit: T-score
Arm/Group | Switch Stable | Treatment-naïve
Number analyzed (Participants) | 2 | 0
T-score
  Femoral Neck Bone Mineral Density: number analyzed (Participants) | 1 | 0
  Femoral Neck Bone Mineral Density | 0.0 [0.0 to 0.0] |
  Lumbar Spine Bone Mineral Density (maximum) | 0.0 [-0.7 to 0.7] |

14. Secondary Outcome: Change From Baseline in Bone Mineral Density (BMD) Assessed by Bone Density Scan (DXA)
Description: An increase in BMD is a positive indicator of efficacy. Subjects had Z-scores reported for change from baseline in Bone Mineral Density in the Femoral Neck and Lumbar Spine regions assessed by Bone Mineral Density (DXA).
  A Z-score compares the subject's bone density to the average bone density of people their own age and gender. If the bones more dense than the average person their own age and gender, the bone mass will be indicated as a positive Z-score. Higher positive Z-score indicates greater bone density. If the bones are less dense than the average person their own age and gender, the bone mass will be indicated as a negative Z-score. Lower negative Z-score indicates lesser bone density.
Time Frame: Baseline to 52 weeks post-AVR-RD-02 treatment follow-up
Population: as for outcome 13
Measure: Mean (Full Range); unit: Z-score
Arm/Group | Switch Stable | Treatment-naïve
Number analyzed (Participants) | 3 | 0
Z-score
  Femoral Neck Bone Mineral Density: number analyzed (Participants) | 2 | 0
  Femoral Neck Bone Mineral Density | 0.45 [0.2 to 0.7] |
  Lumbar Spine Bone Mineral Density | -0.13 [-0.7 to 0.2] |

15. Secondary Outcome: Change From Baseline in Plasma Chitotriosidase Activity Levels Measured by Fluorometric Enzyme Assay
Description: Chitotriosidase enzyme is part of an inflammatory response originating in macrophages, which are the primary cell type affected in Gaucher disease. Gaucher disease patients typically have elevated Chitotriosidase enzyme activity in their plasma compared to healthy population. A reduction from Baseline in chitotriosidase enzyme activity is a positive indicator of efficacy.
Time Frame: Baseline to 52 weeks post-AVR-RD-02 treatment follow-up
Population: Population consists of switch-stable subjects. Treatment-naïve arm do not enroll any subjects at the time of study termination. The secondary efficacy clinical outcome measure was not evaluated as originally planned. (Refer to "Limitations and Caveats" Section.)
Measure: Mean (Full Range); unit: μmol/L/h
Arm/Group | Switch Stable | Treatment-naïve
Number analyzed (Participants) | 2 | 0
μmol/L/h | -37.8 [-70.4 to -5.1] |

16. Secondary Outcome: Change From Baseline in Bone Marrow Burden (BMB) Score as Assessed by Bone Magnetic Resonance Imaging (MRI)
Description: Bone Marrow Burden Score is a semi-quantitative MRI scoring system for assessing the extent of bone marrow involvement in Gaucher disease. A BMB score from 0 to 8 could be given for the lumbar spine, and a BMB score from 0 to 8 could be given to the femurs. Thus, a total BMB score of up to 16 is obtained by adding the lumbar and femoral BMB scores. A higher total BMB-score indicates more severe bone marrow involvement. A reduction in BMB score is a positive indicator of efficacy.
Time Frame: Baseline to 52 weeks post-AVR-RD-02 treatment follow-up
Population: as for outcome 1
Measure: Mean (Full Range); unit: Change from baseline score
Arm/Group | Switch Stable | Treatment-naïve
Number analyzed (Participants) | 4 | 0
Change from baseline score | 0.5 [-1.0 to 1.0] |

ADVERSE EVENTS:
Time Frame: Up to week 52
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience; persistent or significant disability/incapacity; congenital anomaly. The AE/SAE are also inclusive of any abnormalities in Clinical Laboratory Tests, Vital Signs and ECGs.
Groups:
- Switch Stable: Switch-stable arm: Subjects who have undergone ERT ≥15 U/kg and ≤60 U/kg every other week (or equivalent; ie, any combination of infusions resulting in a total monthly ERT dose of >30 U/kg and <120 U/kg) for ≥24 consecutive months for Type 1 Gaucher disease at the time of Screening. Switch-stable subjects must discontinue ERT at least 2 weeks before the scheduled transplant day. Switch-stable subjects who have been on ERT and substrate reduction therapy (SRT) must not have received SRT within 12 months of Screening.
  AVR-RD-02: AVR-RD-02 Drug product: active substance is autologous CD34+ enriched hematopoietic stem cells (HSCs) that have been genetically modified ex vivo with a lentiviral vector (LV) to contain a ribonucleic acid (RNA) transcript that, after reverse transcription, results in codon-optimized, complementary deoxyribonucleic acid (cDNA) that, upon its integration into human genome, encodes for functional human glucocerebrosidase (GCase).
- Treatment-naïve: Treatment-naïve arm: Subjects with Type 1 Gaucher disease who have never received either ERT or SRT for Gaucher disease or have not received either ERT or SRT for Gaucher disease within 12 months of Screening (ie, treatment-naïve subjects). Enrollment will follow a similar scheme as for the switch-stable subjects.
  AVR-RD-02: AVR-RD-02 Drug product: active substance is autologous CD34+ enriched hematopoietic stem cells (HSCs) that have been genetically modified ex vivo with a lentiviral vector (LV) to contain a ribonucleic acid (RNA) transcript that, after reverse transcription, results in codon-optimized, complementary deoxyribonucleic acid (cDNA) that, upon its integration into human genome, encodes for functional human glucocerebrosidase (GCase).
Arm/Group | Switch Stable | Treatment-naïve
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/6 | 0/0
Other Adverse Events (participants affected / at risk) | 6/6 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Switch Stable (N=6) | Treatment-naïve (N=0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Switch Stable (N=6) | Treatment-naïve (N=0)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (5) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (10) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (6) | 0 (0)
Catheter site erythema (General disorders) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0)
Mucosal inflammation (General disorders) | 4 (4) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Swelling (General disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (2) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (2) | 0 (0)
Amylase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0)
B-lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 2 (3) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (2) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 2 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 4 (5) | 0 (0)
Monocyte count decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 5 (8) | 0 (0)
Platelet count decreased (Investigations) | 4 (4) | 0 (0)
Protein total decreased (Investigations) | 1 (1) | 0 (0)
T-lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 5 (6) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Taste disorder (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Azoospermia (Reproductive system and breast disorders) | 1/3 (1) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 1/3 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Red man syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
GCase PBL results were not available at many timepoints due to sample instability. CFB in chitotriosidase was calculated for only 2 subjects because timepoints for the other 2 subjects exceeded ULOQ of the assay and could not be quantified. BMA samples were collected and batched for VCN analysis, but due to study termination, they were not analyzed and thus discarded. Change from baseline BMD scores were not able to be evaluated for some subjects due to missing baseline and/or Week 52 data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT04145037/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-21): https://cdn.clinicaltrials.gov/large-docs/37/NCT04145037/SAP_001.pdf